CLINICAL TRIAL: NCT05292495
Title: A Single-dose, Open Design Study to Evaluate The Pharmacokinetics of HR17031 Injection With Renal Insufficiency
Brief Title: A Trial of HR17031 Injection With Renal Insufficiency
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR17031-105
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Improved Glycemic Control in Patients With Type 2 Diabetes

STUDY DESIGN:
Intervention Model Description: Compare the pharmacokinetics of HR17031 injection in subjects with mild, moderate, severe renal insufficiency and end-stage renal disease and subjects with normal renal function.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort one: mild renal insufficiency (Experimental)
  Interventions: Drug: HR17031 injection
- Cohort two: moderate renal insufficiency (Experimental)
  Interventions: Drug: HR17031 injection
- Cohort three: severe renal insufficiency (Experimental)
  Interventions: Drug: HR17031 injection
- Cohort four: end-stage renal disease (Experimental)
  Interventions: Drug: HR17031 injection
- Cohort five: normal renal function (Experimental)
  Interventions: Drug: HR17031 injection

INTERVENTIONS:
Drug: HR17031 injection — HR17031 injection; administered subcutaneously.

SUMMARY:
This study used a single-dose, open design to compare the pharmacokinetics of subjects with mild, moderate and severe renal insufficiency and end-stage renal disease and subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

- Renal impairment subjects Inclusion Criteria：

1. Signed the informed consent before the test, and fully understood the test content, process and possible adverse reactions; And able to complete the research according to the requirements of the test protocol.
2. Age 18-70 (including threshold), male and female.
3. Body mass index (BMI): 18~30 kg/m2 (including critical value).
4. Creatinine clearance (CLcr, calculated by the Cockcroft-Gault formula) must meet the following criteria:

   Subjects with mild renal insufficiency: 60-89 mL/min (including cutoffs); Subjects with moderate renal impairment: 30-59 mL/min (including cutoffs); Subjects with severe renal impairment: 15-29 mL/min (including cutoffs); Subjects with end-stage renal insufficiency: <15 mL/min.
5. The renal function status is stable, and the CLcr results of the two tests before administration (the two tests need to be separated by at least 3 days, but within 14 days) should be within ±25%. If the second result is not within ±25%, a third test can be performed (at least 3 days from the second test, but within 14 days). The third test result needs to be within ±25% of the second test result. Calculation formula: (third result - second result)/second result. The test results within 24 hours before administration will be used for the final trial grouping and subsequent PK analysis.
6. Females of childbearing age must take reliable contraceptive measures and be willing to use appropriate methods of contraception during the trial and within 10 weeks after the last administration of the test drug; male subjects are willing to have no reproductive plans during the trial and within 10 weeks after the last administration of the test drug and Voluntary use of effective contraception, or surgical sterilization.
7. For patients with other underlying diseases requiring drug treatment, the dose needs to be kept stable during this study.

Healthy subjects Inclusion Criteria：

1. Signed the informed consent before the test, and fully understood the test content, process and possible adverse reactions; And able to complete the research according to the requirements of the test protocol.
2. Able to complete the research in accordance with the requirements of the experimental protocol.
3. Age 18-70 (including threshold), male and female.
4. Body mass index (BMI): 18~30 kg/m2 (including critical value).
5. Creatinine clearance rate (CLcr, calculated by Cockcroft-Gault formula) ≥ 90mL/min.
6. The renal function status is stable, and the CLcr results of the two tests before administration (the two tests need to be separated by at least 3 days, but within 14 days) should be within ±25%. Calculation formula: (second result - first result)/first result. The test results within 24 hours before administration will be used for the final trial grouping and subsequent PK analysis.
7. Females of childbearing age must take reliable contraceptive measures and be willing to use appropriate methods of contraception during the trial and within 10 weeks after the last administration of the test drug; male subjects are willing to have no reproductive plans during the trial and within 10 weeks after the last administration of the test drug and Voluntary use of effective contraception, or surgical sterilization.

Exclusion Criteria:

-

Exclusion Criteria for subjects with mild, moderate and severe renal impairment:

1. Have done kidney transplantation.
2. Renal dialysis is required during the study.
3. Those with allergic constitution, including those with a history of severe drug allergy or drug allergy, or known or suspected to be allergic to any component in the study drug.
4. Urinary incontinence or anuria (eg <100ml/d).
5. Those who have a history of drug and/or alcohol abuse, who are positive for alcohol and drug screening, or who have a history of drug abuse in the past five years or who have used drugs in the 3 months before the test; and who cannot smoke or abstain from alcohol during the test.
6. Pregnant or lactating women, or those with a positive blood pregnancy result.
7. Those who donated blood or participated in any clinical trial drugs within 3 months before screening.
8. Those who have taken other prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplements other than those used to treat renal insufficiency and other concomitant diseases within 14 days before administration.
9. Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive or combined with positive syphilis serology).
10. Major surgery or surgical incision was not fully healed within 6 months before screening.
11. History or clinical symptoms of deep vein thrombosis or other thromboembolic events suggest thrombophilia.
12. Active heart disease within 6 months before the first administration of the study drug, including: severe/unstable angina pectoris, myocardial infarction, symptomatic congestive heart failure and ventricular arrhythmia requiring drug treatment.
13. Have a history of epilepsy, or a disease that can induce epileptic seizures within 12 months before the first administration of the study drug (including a history of transient ischemic attack, cerebral apoplexy (except for cerebral ischemic lesions found by simple imaging examination), Brain trauma with disturbance of consciousness requires hospitalization).
14. Malignant tumors, or a history of malignant tumors within 5 years before screening (except for skin non-melanoma that has been treated and has no signs of recurrence, and excised cervical intraepithelial neoplasia).
15. In addition to renal insufficiency and other concomitant diseases, the researcher makes judgments based on medical history inquiry, comprehensive physical examination, routine laboratory tests (blood routine, blood biochemistry, urine routine, etc.), X-chest X-ray, abdominal B-ultrasound, etc. Abnormal clinical significance.

16、12-ECG abnormality with clinical significance and uncontrollable by drugs (if uncontrolled tachycardia/bradycardia, II-III degree atrioventricular block or prolongation of QTcF interval (male ≥ 470 ms, female ≥ 470 ms) 480 ms) (corrected by Fridericia's formula) or other clinically significant abnormalities judged by the clinician).

17、48 hours before taking the study drug until the end of the study, the subject refuses to stop any beverages containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, etc.) or alcoholic beverages or any fruit juice.

18、Vigorous exercise within 48 hours before administration, or other factors affecting drug distribution, metabolism, excretion, etc..

19、Those with a history of fainting, fainting of blood, difficult to collect blood or unable to tolerate venipuncture for blood collection.

20、Those who have used insulin or glucagon-like polypeptide-1 receptor agonist (GLP-1) hypoglycemic drugs within 3 months before screening.

21、Those who have been vaccinated or exposed to other live vaccines or live attenuated vaccines within 3 months before screening; or those who plan to receive live vaccines or live attenuated vaccines during the study period.

22、According to the judgment of the researcher, there are concomitant diseases (such as poorly controlled hypertension, severe diabetes, thyroid disease and mental illness, etc.) or any other conditions that seriously endanger the safety of patients, or affect the completion of the study.

Exclusion Criteria for ESRD:

1. Have done kidney transplantation.
2. Those with allergic constitution, including those with a history of severe drug allergy or drug allergy, or known or suspected to be allergic to any component of the study drug.
3. Urinary incontinence or anuria (eg <100ml/d).
4. Those who have a history of drug and/or alcohol abuse, who are positive for alcohol and drug screening, or who have a history of drug abuse in the past five years or who have used drugs in the 3 months before the test; and who cannot smoke and abstain during the test.
5. Pregnant or lactating women, or those with a positive blood pregnancy result.
6. Those who donated blood or participated in any clinical trial drug within 3 months before screening.
7. Those who have taken other prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplements other than those used to treat renal insufficiency and other concomitant diseases within 14 days before administration.
8. Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive or combined with positive syphilis serology).
9. Received major surgery within 6 months before screening or the surgical incision was not completely healed.
10. History or clinical symptoms of deep vein thrombosis or other thromboembolic events suggest thrombophilia.
11. Active heart disease within 6 months before the first administration of the study drug, including: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure and ventricular arrhythmia requiring drug treatment.
12. Have a history of epilepsy, or a disease that can induce epileptic seizures within 12 months before the first administration of the study drug (including a history of transient ischemic attack, cerebral apoplexy (except for cerebral ischemic lesions found by simple imaging examination), Brain trauma with disturbance of consciousness requires hospitalization).
13. Suffering from malignant tumor, or a history of malignant tumor within 5 years before screening (except for skin non-melanoma that has been treated and has no signs of recurrence, and excised cervical intraepithelial neoplasia).
14. In addition to renal insufficiency and other concomitant diseases, the researcher makes judgments based on medical history inquiry, comprehensive physical examination, routine laboratory tests (blood routine, blood biochemistry, urine routine, etc.), X-chest X-ray, abdominal B-ultrasound, etc. Abnormal clinical significance.

    15、12-ECG abnormality is clinically significant and uncontrollable by drugs (if uncontrolled tachycardia/bradycardia, II-III degree atrioventricular block or prolongation of QTcF interval (men ≥ 470 ms, women ≥ 470 ms) 480 ms) (corrected by Fridericia's formula) or other clinically significant abnormalities judged by the clinician).

    16、48 hours before taking the study drug until the end of the study, the subject refuses to stop any beverages containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, etc.) or alcoholic beverages or any fruit juice.

17、Vigorous exercise within 48 hours before administration, or other factors affecting drug distribution, metabolism, excretion, etc..

18、Those with a history of fainting of needles, fainting of blood, difficulty in blood collection or intolerance of venipuncture for blood collection.

19、Those who have used insulin or glucagon-like polypeptide-1 receptor agonist (GLP-1) hypoglycemic drugs within 3 months before screening.

20、Those who have been vaccinated or exposed to other live vaccines or live attenuated vaccines within 3 months before screening; or those who plan to receive live vaccines or live attenuated vaccines during the study period.

21、According to the judgment of the researcher, there are concomitant diseases (such as poorly controlled hypertension, severe diabetes, thyroid disease and mental illness, etc.) or any other conditions that seriously endanger the safety of patients, or affect the completion of the study.

Exclusion Criteria for Healthy subject:

1. Chronic kidney disease damage and kidney transplantation.
2. Those with allergic constitution, including those with a history of severe drug allergy or drug allergy, or known or suspected to be allergic to any component of the study drug.
3. Those who have a history of drug and/or alcohol abuse, who are positive for alcohol and drug screening, or who have a history of drug abuse in the past five years or who have used drugs in the 3 months before the test; and who cannot smoke or abstain from alcohol during the test.
4. Pregnant or breastfeeding women, or those with a positive blood pregnancy result.
5. Those who donated blood or took any clinical trial drugs within 3 months before screening.
6. Those who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplements within 14 days before administration.
7. Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive or combined with positive syphilis serology).
8. Those who have undergone any surgery within 6 months before screening.
9. History or clinical symptoms of deep vein thrombosis or other thromboembolic events suggest thrombophilia.
10. Active heart disease within 6 months before the first administration of the study drug, including: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure and ventricular arrhythmia requiring drug treatment.
11. Have a history of epilepsy, or a disease that can induce epileptic seizures within 12 months before the first administration of the study drug (including history of transient ischemic attack, cerebral apoplexy (except for cerebral ischemic foci found by simple imaging examination), Brain trauma with disturbance of consciousness requires hospitalization).
12. Suffering from malignant tumor, or a history of malignant tumor within 5 years before screening (except for skin non-melanoma that has been treated and has no signs of recurrence, and excised cervical intraepithelial neoplasia).
13. Comprehensive physical examination (vital signs, physical examination), routine laboratory examinations (blood routine, blood biochemistry, urine routine, thrombin function, etc.), X-chest X-ray, abdominal B-ultrasound and other abnormal examinations with clinical significance.

14、12-ECG abnormalities with clinical significance and uncontrollable by drugs (if uncontrolled tachycardia/bradycardia, II-III degree atrioventricular block or prolongation of QTcF interval (≥470 ms in males, ≥470 ms in females) 480 ms) (corrected by Fridericia's formula) or other clinically significant abnormalities judged by the clinician).

15、48 hours before taking the study drug until the end of the study, the subject refuses to stop any beverages containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, etc.) or alcoholic beverages or any fruit juice.

16、Vigorous exercise within 48 hours before administration, or other factors affecting drug distribution, metabolism, excretion, etc..

17、Those with a history of needle fainting, haemorrhage, difficulty in blood collection or intolerance of venipuncture for blood collection.

18、Those who have used insulin or glucagon-like polypeptide-1 receptor agonist (GLP-1) hypoglycemic drugs within 3 months before screening.

19、Those who have been vaccinated or exposed to other live vaccines or live attenuated vaccines within 3 months before screening; or those who plan to receive live vaccines or live attenuated vaccines during the study period.

20、According to the judgment of the investigator, there are concomitant diseases (such as poorly controlled hypertension, severe diabetes, thyroid disease and mental illness, etc.) or any other conditions that seriously endanger the safety of patients, or affect the completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-03-31 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of INS068 and SHR20004: Cmax | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: AUC0-t | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: AUC0-inf | Based on pre-dose, 2-96 hours post-dose sampling times

SECONDARY OUTCOMES:
Pharmacokinetics parameters of INS068 and SHR20004: Tmax | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: T1/2 | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: CL/F | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: Vz/F | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: Ae | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: fe | Based on pre-dose, 2-96 hours post-dose sampling times
Pharmacokinetics parameters of INS068 and SHR20004: CLr | Based on pre-dose, 2-96 hours post-dose sampling times
Average concentrations of INS068 and SHR20004 in dialysate of ESRD | 0- 4 hours post-dose sampling times
Cumulative collection amount of INS068 and SHR20004 in dialysate of ESRD | 0- 4 hours post-dose sampling times
Dialysis clearance of INS068 and SHR20004 in dialysate of ESRD | 0- 4 hours post-dose sampling times
Binding rate of plasma protein of INS068 in serum and SHR20004 in plasma(fu) | Based on pre-dose, 2-96 hours post-dose sampling times
The incidence and severity of adverse events/serious adverse events | Based on pre-dose, 2-96 hours post-dose sampling times
ADA：anti-drug antibody | Based on pre-dose、Day 5、Day14、Day 24 or early termination

IPD SHARING:
Plan to Share IPD: Undecided